CLINICAL TRIAL: NCT02358005
Title: Optimal Dose of Extracorporeal Shock Wave Therapy After Botulinum Toxin Type A Injection for Post-stroke Spasticity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2014-0925
Record Dates: First submitted 2015-01-23; First posted 2015-02-06 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Post-Stroke Elbow Spasticity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 60mJ ESWT (Experimental): ESWT (0.04 mJ/mm2, 1500 shock + sham stimulation 2500) / total dose per treatment : 60mJ
  Interventions: Procedure: Extracorporeal shock wave therapy 60mj
- 120mJ ESWT (Experimental): ESWT (0.04 mJ/mm2, 4000 shock) / total dose per treatment : 160mJ
  Interventions: Procedure: Extracorporeal shock wave therapy 120mj
- sham ESWT stimulation (Placebo Comparator): ESWT (0 mJ/mm2, sham stimulation 4000) / total dose per treatment : 0mJ
  Interventions: Procedure: non extracorporeal shock wave therapy

INTERVENTIONS:
Procedure: Extracorporeal shock wave therapy 60mj
  Arms: 60mJ ESWT
Procedure: Extracorporeal shock wave therapy 120mj
  Arms: 120mJ ESWT
Procedure: non extracorporeal shock wave therapy
  Arms: sham ESWT stimulation

SUMMARY:
Recently, It is known that the efficacy of botulinum toxin type A (BTX-A) with extracorporeal shock wave therapy (ESWT) is greater than that of BTX-A with electrical stimulation in the management of post-stroke spasticity of the upper limb. However, it was not determined which dose of ESWT is optimal as a adjuvant therapy after BTX-A injection on the upper limb in patients with stroke. Therefore, the aim of this study is to evaluate the optimal dose of ESWT after botulinum toxin type A injection for post-stroke spasticity

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥20 years
* inpatients
* Elbow flexor spasticity in patients, confirmed to be mainly due to biceps brachii
* Modified Ashworth scale (MAS) ≥2,
* At least a 3-month period from stroke,
* Written informed consent has been obtained

Exclusion Criteria:

* Fixed contractures and/or deformities at the elbow,
* Previous fractures of the paretic upper limb,
* Peripheral nervous system disorders/myopathies,
* Previous BTX-A treatment and/or ESWT,
* Structural alterations in the soft tissue (e.g., fibrosis),
* Known allergy or sensitivity to the study medication or its components
* Presence of an unstable medical condition or uncontrolled systemic disease
* Any medical condition that may put the patient at increased risk with exposure to botulinum toxin therapy. (ex. Myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interface with neuromuscular function.
* Bleeding tendency and/or anticoagulation therapy
* Presence of infection or skin disorder at injection sites
* Females were are pregnant, nursing, or are planning a pregnancy during the study
* Females of child-bearing potential (including pre-menstrual woman), not using a reliable means of contraception
* Participant who should be withdrawn from the study in the opinion of the investigator for any reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Range of Motion (ROM) of elbow flexor | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Healthcare System, Severance Hospital, Seoul, South Korea